CLINICAL TRIAL: NCT05585255
Title: Clinical Significance, Mechanism of Action, and New Targeted Drug Research of DKK2 Protein in Cerebral Ischemia-reperfusion Injury
Brief Title: Clinical Significance of DKK2 Protein in Cerebral Ischemia-reperfusion Injury
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huang Kaibin, associate chief physician, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2022-273
Record Dates: First submitted 2022-09-21; First posted 2022-10-18 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke, Acute; Ischemia-reperfusion Injury; Cerebral Edema
MeSH Terms: conditions — Ischemic Stroke; Reperfusion Injury; Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Venous blood samples of acute stroke patients with revascularisation treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke patients: Acute ischemic stroke patients with large vessel occlusion who received mechanical thrombectomy therapy and are successfully revascularized
  Interventions: Diagnostic Test: enzyme-linked immunosorbent assay(ELISA)

INTERVENTIONS:
Diagnostic Test: enzyme-linked immunosorbent assay(ELISA) — After allowing to stand at room temperature for 2h, blood samples are centrifuged at 4 ℃ for 15 min (12000 rpm) to collect the supernatant. Then, the levels of DKK2, IL-6, IL-1β, TNF-α, and IL-10 in the supernatants are tested by ELISA detection.

SUMMARY:
The study is a two-center prospective cohort clinical trial. The primary purpose of this trial is to identify the pattern of DKK2 serum levels in ischemic stroke patients after revascularization therapy and determine the correlation between serum DKK2 levels and prognosis.

DETAILED DESCRIPTION:
Ischemic stroke refers to ischaemic and hypoxic necrosis of brain tissue caused by narrowing or occlusion of the blood vessels in the brain and accounts for approximately 80% of all strokes. It is characterized by high morbidity, mortality, disability, and recurrence rates. Reperfusion is currently the most effective treatment for the acute phase of ischaemic stroke, including pharmacological thrombolysis and mechanical embolization. Although successful revascularization can reperfuse areas of cerebral ischemia, it can cause acute cerebrovascular damage while restoring blood supply to brain tissue, leading to disruption of the blood-brain barrier (BBB), increased risk of cerebral edema and hemorrhagic transformation, and increased inflammation of neural tissue, which can further damage brain tissue. Targeted reduction of endothelial damage from ischemia-reperfusion will therefore effectively protect neurons from subsequent damage, thereby minimizing neurological impairment after stroke and maximizing the benefit of revascularisation therapy.

The Wnt signaling pathway has been identified by several research groups worldwide as a key regulatory pathway in the maintenance of cerebrovascular and neural cell function. The DKK (Dickkopf-related protein) family of proteins is the most representative group of classical Wnt signaling pathway inhibitors. DKK proteins competitively bind to the Wnt co-receptor LRP5/6, thereby inhibiting the activity of Wnt proteins and exerting their inhibitory effects on the Wnt/β-catenin signaling pathway. We initially found that DKK2 serum levels increased significantly after 4.5 h of recanalization therapy in 20 patients with large vessel occlusive acute stroke, and decreased after 24 h. Increased DKK2 levels were strongly associated with an unfavorable prognosis. This was corroborated in animal models as well, DKK2 expression levels in ischaemic brain tissue and peripheral blood were both significantly elevated and rapidly upregulated within 6-12 h of the onset of cerebral ischemia-reperfusion in mice. In vitro cellular assays showed that DKK2 protein significantly inhibited the activity of the Wnt/β-catenin signaling pathway. We further study showed that upregulation of DKK2 protein levels in the blood of mice by intravenous administration of adenovirus expressing DKK2 protein significantly increased cerebral infarction and neurological impairment in mice with stroke. The increased expression of DKK2 protein in brain tissue is the main reason for the downregulation of Wnt/β-catenin signaling pathway activity after ischemia/reperfusion, which leads to blood-brain barrier damage, neuronal cell death, and neuroinflammation, and ultimately promotes brain tissue damage and neurological dysfunction. It is a new target for drug therapy and has great scientific significance and clinical application prospects.

This clinical study is conducted at Dongguan Hospital of Southern Medical University and Nanfang Hospital of Southern Medical University. Acute ischemic stroke patients with large vessel occlusion who received mechanical thrombectomy therapy and are successfully revascularized will be included and followed up for 90 d, along with testing serum levels of DKK2 protein to explore its correlation with the prognosis of enrolled patients. Venous blood samples will be collected before, and 24 h, 48 h, and 72 h after revascularization treatment in enrolled patients. Venous blood samples will be collected before and 0h, 24 h, 48 h, and 72 h after revascularisation treatment to test serum KKD2 level, and cranial CT examination will be performed before, 24 h, and 72 h after revascularization treatment to detect the occurrence of the transformation of hemorrhage, the severity of cerebral edema, and midline shift after revascularisation treatment. Blood-brain barrier injury-related indicators (MMP-9, ICAM-1) and inflammation-related indicators (IL-6, IL-1β, TNF-α, IL-10) will be measured at each time point of DKK2 testing. NIHSS scores will be evaluated before, 0h (immediately after revascularization treatment), 24 h, 48 h, 72 h, and 7 d after revascularization treatment. The mRS scores will be followed up at 30 days and 90 days after the onset to clarify the relationship between serum DKK2 levels and large vessel occlusion. We aim to investigate the mechanism of DKK2 causing adverse clinical outcomes such as BBB leakage, cerebral edema, and hemorrhagic transformation at a real-world clinical level by collecting blood samples, clinical follow-up, and neurological scoring from stroke patients by measuring DKK2 levels and brain imaging parameters for quantitative assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, < 80 years, sex not limited;
2. Definite clinical diagnosis of acute ischemic stroke;
3. Baseline NIHSS score ≥ 6 and ≤ 25;
4. CTA/MRA/DSA examination suggests large vessel occlusion in the anterior circulation (internal carotid artery, M1/M2 segment of the middle cerebral artery);
5. The criteria for receiving endovascular treatment in accordance with the Chinese Guidelines for Early Endovascular Intervention in Acute Ischemic Stroke 2018 and have successful revascularization (TICI ≥ grade 2b);
6. Subjects or their legal representatives agree to the treatment and sign the informed consent form.

Exclusion Criteria:

1. Patients with combined posterior circulation infarction;
2. The mRS ≥ 2 points before the current episode;
3. Patients who are to be treated with or have been treated with anticoagulants;
4. Patients with existing or active organ bleeding within 6 months of enrollment, including cerebral hemorrhage, subarachnoid hemorrhage, gastrointestinal tract hemorrhage, fundus hemorrhage, etc;
5. The presence of other intracranial pathologies, such as cerebrovascular malformations, cerebral venous lesions, tumors, and other diseases involving the cranium;
6. Severe organ dysfunction or failure;
7. Those with severe hematologic disorders or severe coagulation abnormalities；
8. Those with a history of severe trauma or major surgical procedures within 6 months prior to enrollment;
9. Pregnant or lactating women;
10. Patients with a life expectancy of less than 3 months or who for other reasons are unable to complete the study;
11. Unwillingness to be followed up or poor compliance with treatment;
12. Other conditions that the investigator considers unsuitable for enrollment.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients with large vessel occlusion who are treated with mechanical embolization and successfully revascularized at Dongguan Hospital of Southern Medical University and Nanfang Hospital of Southern Medical University.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
90-day Functional Outcome. | The mRS score will follow up at 90 days.
  The favorable prognosis (modified Rankin score [mRS] score ≤ 2) and the unfavorable prognosis group ([mRS] score ≥ 3) within 90 d after onset.

SECONDARY OUTCOMES:
Incidence of neurological deterioration | The NIHSS score will evaluat at the point before revascularization treatment, 0 (immediately after revascularization treatment), 24, 48, 72 hours, and 7 days after revascularization treatment.
  Significantly improved NIHSS score (an increase in the NIHSS score by ≥4 points) within 7 days after onset.
Incidence of substantial hemorrhagic transformation | At the point before revascularization treatment, 24, and 72 hours after revascularization treatment.
  Cranial CT examination will perform to detect substantial hemorrhagic transformation (ECASS typing PH2 type) within 72 hours.
The severity of cerebral edema. | At the point before revascularization treatment, 24, and 72 hours after revascularization treatment.
  Cranial CT examination will perform to detect the varying severity of cerebral edema groups (divided into 3 groups according to CED scores 1, 2 and 3) within 72 hours.
Incidence of midline shift ≥ 6mm. | At the point before revascularization treatment, 24, and 72 hours after revascularization treatment.
  Cranial CT examination will perform to detect the severity of cerebral edema and cerebral hernia.
Levels of major inflammatory indicators in peripheral blood. | Before revascularization treatment, 24, 48, 72 hours and 7 days after revascularization treatment.
  Blood-brain barrier injury-related indicators (MMP-9, ICAM-1) and inflammation-related indicators (IL-6, IL-1β, TNF-α, IL-10).

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Shi, PHD, Study Chair — Dongguan Hospital of Southern Medical University
Locations (2):
- China (2):
  - Dongguan Hospital of Southern Medical University, Dongguan, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.

REFERENCES:
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Phipps MS, Cronin CA. Management of acute ischemic stroke. BMJ. 2020 Feb 13;368:l6983. doi: 10.1136/bmj.l6983. PMID 32054610
- [Background] Ma H, Campbell BCV, Parsons MW, Churilov L, Levi CR, Hsu C, Kleinig TJ, Wijeratne T, Curtze S, Dewey HM, Miteff F, Tsai CH, Lee JT, Phan TG, Mahant N, Sun MC, Krause M, Sturm J, Grimley R, Chen CH, Hu CJ, Wong AA, Field D, Sun Y, Barber PA, Sabet A, Jannes J, Jeng JS, Clissold B, Markus R, Lin CH, Lien LM, Bladin CF, Christensen S, Yassi N, Sharma G, Bivard A, Desmond PM, Yan B, Mitchell PJ, Thijs V, Carey L, Meretoja A, Davis SM, Donnan GA; EXTEND Investigators. Thrombolysis Guided by Perfusion Imaging up to 9 Hours after Onset of Stroke. N Engl J Med. 2019 May 9;380(19):1795-1803. doi: 10.1056/NEJMoa1813046. PMID 31067369
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Patel P, Yavagal D, Khandelwal P. Hyperacute Management of Ischemic Strokes: JACC Focus Seminar. J Am Coll Cardiol. 2020 Apr 21;75(15):1844-1856. doi: 10.1016/j.jacc.2020.03.006. PMID 32299596
- [Background] Yang P, Zhang Y, Zhang L, Zhang Y, Treurniet KM, Chen W, Peng Y, Han H, Wang J, Wang S, Yin C, Liu S, Wang P, Fang Q, Shi H, Yang J, Wen C, Li C, Jiang C, Sun J, Yue X, Lou M, Zhang M, Shu H, Sun D, Liang H, Li T, Guo F, Ke K, Yuan H, Wang G, Yang W, Shi H, Li T, Li Z, Xing P, Zhang P, Zhou Y, Wang H, Xu Y, Huang Q, Wu T, Zhao R, Li Q, Fang Y, Wang L, Lu J, Li Y, Fu J, Zhong X, Wang Y, Wang L, Goyal M, Dippel DWJ, Hong B, Deng B, Roos YBWEM, Majoie CBLM, Liu J; DIRECT-MT Investigators. Endovascular Thrombectomy with or without Intravenous Alteplase in Acute Stroke. N Engl J Med. 2020 May 21;382(21):1981-1993. doi: 10.1056/NEJMoa2001123. Epub 2020 May 6. PMID 32374959
- [Background] Moskowitz MA, Lo EH, Iadecola C. The science of stroke: mechanisms in search of treatments. Neuron. 2010 Jul 29;67(2):181-98. doi: 10.1016/j.neuron.2010.07.002. PMID 20670828
- [Background] Shi K, Zou M, Jia DM, Shi S, Yang X, Liu Q, Dong JF, Sheth KN, Wang X, Shi FD. tPA Mobilizes Immune Cells That Exacerbate Hemorrhagic Transformation in Stroke. Circ Res. 2021 Jan 8;128(1):62-75. doi: 10.1161/CIRCRESAHA.120.317596. Epub 2020 Oct 19. PMID 33070717
- [Background] Wang R, Zhu Y, Liu Z, Chang L, Bai X, Kang L, Cao Y, Yang X, Yu H, Shi MJ, Hu Y, Fan W, Zhao BQ. Neutrophil extracellular traps promote tPA-induced brain hemorrhage via cGAS in mice with stroke. Blood. 2021 Jul 8;138(1):91-103. doi: 10.1182/blood.2020008913. PMID 33881503
- [Background] El-Benna J, Hurtado-Nedelec M, Marzaioli V, Marie JC, Gougerot-Pocidalo MA, Dang PM. Priming of the neutrophil respiratory burst: role in host defense and inflammation. Immunol Rev. 2016 Sep;273(1):180-93. doi: 10.1111/imr.12447. PMID 27558335
- [Background] Chen R, Zhang X, Gu L, Zhu H, Zhong Y, Ye Y, Xiong X, Jian Z. New Insight Into Neutrophils: A Potential Therapeutic Target for Cerebral Ischemia. Front Immunol. 2021 Jul 14;12:692061. doi: 10.3389/fimmu.2021.692061. eCollection 2021. PMID 34335600
- [Background] Jian Z, Liu R, Zhu X, Smerin D, Zhong Y, Gu L, Fang W, Xiong X. The Involvement and Therapy Target of Immune Cells After Ischemic Stroke. Front Immunol. 2019 Sep 11;10:2167. doi: 10.3389/fimmu.2019.02167. eCollection 2019. PMID 31572378
- [Background] O'Collins VE, Macleod MR, Donnan GA, Horky LL, van der Worp BH, Howells DW. 1,026 experimental treatments in acute stroke. Ann Neurol. 2006 Mar;59(3):467-77. doi: 10.1002/ana.20741. PMID 16453316
- [Background] Zhou Z, Lu J, Liu WW, Manaenko A, Hou X, Mei Q, Huang JL, Tang J, Zhang JH, Yao H, Hu Q. Advances in stroke pharmacology. Pharmacol Ther. 2018 Nov;191:23-42. doi: 10.1016/j.pharmthera.2018.05.012. Epub 2018 May 25. PMID 29807056
- [Background] Elkins J, Veltkamp R, Montaner J, Johnston SC, Singhal AB, Becker K, Lansberg MG, Tang W, Chang I, Muralidharan K, Gheuens S, Mehta L, Elkind MSV. Safety and efficacy of natalizumab in patients with acute ischaemic stroke (ACTION): a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Neurol. 2017 Mar;16(3):217-226. doi: 10.1016/S1474-4422(16)30357-X. Epub 2017 Feb 15. PMID 28229893
- [Background] Nusse R, Clevers H. Wnt/beta-Catenin Signaling, Disease, and Emerging Therapeutic Modalities. Cell. 2017 Jun 1;169(6):985-999. doi: 10.1016/j.cell.2017.05.016. PMID 28575679
- [Background] Clevers H, Nusse R. Wnt/beta-catenin signaling and disease. Cell. 2012 Jun 8;149(6):1192-205. doi: 10.1016/j.cell.2012.05.012. PMID 22682243
- [Background] Routledge D, Scholpp S. Mechanisms of intercellular Wnt transport. Development. 2019 May 15;146(10):dev176073. doi: 10.1242/dev.176073. PMID 31092504
- [Background] Chang J, Mancuso MR, Maier C, Liang X, Yuki K, Yang L, Kwong JW, Wang J, Rao V, Vallon M, Kosinski C, Zhang JJ, Mah AT, Xu L, Li L, Gholamin S, Reyes TF, Li R, Kuhnert F, Han X, Yuan J, Chiou SH, Brettman AD, Daly L, Corney DC, Cheshier SH, Shortliffe LD, Wu X, Snyder M, Chan P, Giffard RG, Chang HY, Andreasson K, Kuo CJ. Gpr124 is essential for blood-brain barrier integrity in central nervous system disease. Nat Med. 2017 Apr;23(4):450-460. doi: 10.1038/nm.4309. Epub 2017 Mar 13. PMID 28288111
- [Background] Ji YB, Gao Q, Tan XX, Huang XW, Ma YZ, Fang C, Wang SN, Qiu LH, Cheng YX, Guo FY, Chang J. Lithium alleviates blood-brain barrier breakdown after cerebral ischemia and reperfusion by upregulating endothelial Wnt/beta-catenin signaling in mice. Neuropharmacology. 2021 Mar 15;186:108474. doi: 10.1016/j.neuropharm.2021.108474. Epub 2021 Jan 29. PMID 33524408
- [Background] Ta S, Rong X, Guo ZN, Jin H, Zhang P, Li F, Li Z, Lin L, Zheng C, Gu Q, Zhang Y, Liu W, Yang Y, Chang J. Variants of WNT7A and GPR124 are associated with hemorrhagic transformation following intravenous thrombolysis in ischemic stroke. CNS Neurosci Ther. 2021 Jan;27(1):71-81. doi: 10.1111/cns.13457. Epub 2020 Sep 29. PMID 32991049
- [Background] Song D, Zhang X, Chen J, Liu X, Xue J, Zhang L, Lan X. Wnt canonical pathway activator TWS119 drives microglial anti-inflammatory activation and facilitates neurological recovery following experimental stroke. J Neuroinflammation. 2019 Dec 6;16(1):256. doi: 10.1186/s12974-019-1660-8. PMID 31810470
- [Background] Wei ZZ, Zhang JY, Taylor TM, Gu X, Zhao Y, Wei L. Neuroprotective and regenerative roles of intranasal Wnt-3a administration after focal ischemic stroke in mice. J Cereb Blood Flow Metab. 2018 Mar;38(3):404-421. doi: 10.1177/0271678X17702669. Epub 2017 Apr 21. PMID 28430000
- [Background] Wang W, Li M, Wang Y, Wang Z, Zhang W, Guan F, Chen Q, Wang J. GSK-3beta as a target for protection against transient cerebral ischemia. Int J Med Sci. 2017 Mar 11;14(4):333-339. doi: 10.7150/ijms.17514. eCollection 2017. PMID 28553165
- [Background] Wu MV, Hen R. The young and the restless: regulation of adult neurogenesis by Wnt signaling. Cell Stem Cell. 2013 Feb 7;12(2):139-40. doi: 10.1016/j.stem.2013.01.013. PMID 23395437
- [Background] Busceti CL, Biagioni F, Aronica E, Riozzi B, Storto M, Battaglia G, Giorgi FS, Gradini R, Fornai F, Caricasole A, Nicoletti F, Bruno V. Induction of the Wnt inhibitor, Dickkopf-1, is associated with neurodegeneration related to temporal lobe epilepsy. Epilepsia. 2007 Apr;48(4):694-705. doi: 10.1111/j.1528-1167.2007.01055.x. PMID 17437412
- [Background] Cappuccio I, Calderone A, Busceti CL, Biagioni F, Pontarelli F, Bruno V, Storto M, Terstappen GT, Gaviraghi G, Fornai F, Battaglia G, Melchiorri D, Zukin RS, Nicoletti F, Caricasole A. Induction of Dickkopf-1, a negative modulator of the Wnt pathway, is required for the development of ischemic neuronal death. J Neurosci. 2005 Mar 9;25(10):2647-57. doi: 10.1523/JNEUROSCI.5230-04.2005. PMID 15758175
- [Background] Mastroiacovo F, Busceti CL, Biagioni F, Moyanova SG, Meisler MH, Battaglia G, Caricasole A, Bruno V, Nicoletti F. Induction of the Wnt antagonist, Dickkopf-1, contributes to the development of neuronal death in models of brain focal ischemia. J Cereb Blood Flow Metab. 2009 Feb;29(2):264-76. doi: 10.1038/jcbfm.2008.111. Epub 2008 Oct 1. PMID 18827832